CLINICAL TRIAL: NCT07231003
Title: The Effect of Glucomannan Powder on Improving Gut Microbiota.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: lin5611_03
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dysbiosis
Keywords: dysbiosis; Glucomannan; gut-microbiota
MeSH Terms: conditions — Dysbiosis | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): 2 packs of corn starch daily
  Interventions: Dietary Supplement: Placebo
- Intervention group (Experimental): 2 packs of glucomannan powder daily
  Interventions: Dietary Supplement: Glucomannan

INTERVENTIONS:
Dietary Supplement: Glucomannan — 2 packs of glucomannan, 2 grams per pack
  Arms: Intervention group
Dietary Supplement: Placebo — 2 packs of corn starch, 2 grams per pack
  Arms: Placebo group

SUMMARY:
The object of this study is evaluating the effects of the Glucommanan on the healthy human subjects who are. In this trial, at most 30 healthy subjects whose ages are 20~65 years old (15 for placebo and 15 for intervention)will be included. The total experiment will be 9 weeks and the intervention period will be 6 weeks, within which, at week 0, 6, and 7, total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), aspartate aminotransferase (AST, also known as GOT), alanine aminotransferase (ALT, also known as GPT), blood urea nitrogen (BUN), serum creatinine (Cr), fasting blood glucose (Glucose, AC) and adiponectin would be measured. Feces samples and anthropometric data will also be acquired. The results will be analyzed according to the methods published by the Ministry of Health and Welfare of Taiwan Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

- Both genders, aged between 20 and 65 years.

No history of gastrointestinal disorders or other significant health issues.

Overall good health.

Exclusion Criteria:

- Participants who have taken antibiotics or any medications/supplements that could affect the gut microbiota within 1 week prior to the experiment or during the study.

Pregnant or breastfeeding women.

Smokers or individuals with excessive alcohol consumption.

Chronic disease medication usage for less than 3 months.

Postmenopausal women on hormone replacement therapy.

Individuals with acute illnesses such as a cold.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
gut microbiota | Week(0) (Baseline), Wk(6),Wk7
  Evaluation of Gut Microbiota by Analysis of Four Indicator Strains and 16S rRNA Sequencing Using Fecal Samples

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided